CLINICAL TRIAL: NCT06977932
Title: The Alternative Effects of Electroacupuncture in the Treatment of Trigeminal Neuralgia: Protocol for a Multicentre Randomised Controlled Trial
Brief Title: The Alternative Effects of Electroacupuncture in the Treatment of Trigeminal Neuralgia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yuanyuan Wu (Other)
Collaborators: Pingyang County Traditional Chinese Medicine Hospital (Unknown); Jiaxing Traditional Chinese Medicine Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Yuanyuan Wu, Associate Professor, The Third Affiliated hospital of Zhejiang Chinese Medical University
Organization: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GZY-KJS-ZJ-2025-006-ALT
Record Dates: First submitted 2025-05-11; First posted 2025-05-18 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Trigeminal Neuralgia
Keywords: Electroacupuncture; Randomized Controlled Trial
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sham EA +CBZ group (Sham Comparator): A cohort of 63 patients with TN will undergo treatment with CBZ in conjunction with a sham EA intervention.
  Interventions: Drug: Carbarmazepine; Procedure: Sham Electroacupuncture
- EA+placebo group (Experimental): A cohort of 63 patients diagnosed with TN will undergo treatment involving a combination of placebo and EA. The EA procedures will be administered by licensed acupuncturists who have received standardized training.
  Interventions: Drug: Carbarmazepine Placebo; Procedure: Electroacupuncture

INTERVENTIONS:
Drug: Carbarmazepine — Following enrollment, the patient's carbamazepine dosage remained consistent with the pre-enrollment dosage. Orally administered for two consecutive weeks.
  Arms: sham EA +CBZ group
Procedure: Sham Electroacupuncture — In this group, superficial needling (0.5-1 mm depth) was performed at non-meridian points located 1 cm lateral to: (1) primary local acupoints ST2 (Sibai), ST7 (Xiaguan), and ST4 (Dicang) on the affected side; (2) branch-specific supplementary points GB1 (Tongziliao) for ophthalmic branch involvement, SI18 (Quanliao) for maxillary branch involvement, and ST6 (Jiache) for mandibular branch involvement; and (3) bilateral distal points LI4 (Hegu) and TE5 (Waiguan). Local acupoint pairs (ST7 adjacent + GB1 adjacent, ST7 adjacent + SI18 adjacent, or ST7 adjacent + ST6 adjacent) and distal pairs (LI4 adjacent + TE5 adjacent) were connected to an electroacupuncture device. The electroacupuncture device was kept in the off state and did not generate any therapeutic current. The needles were retained for 60 minutes.Acupuncture treatment was administered for 5 consecutive days as one course, with a 2-day break between courses. A total of 2 courses were conducted.
  Arms: sham EA +CBZ group
Drug: Carbarmazepine Placebo — CBZ placebo is a tablet with identical packaging and appearance to CBZ but lacks therapeutic effects. Patients were transitioned to a CBZ placebo at an equivalent daily dose post-enrollment. Orally administered for two consecutive weeks.
  Arms: EA+placebo group
Procedure: Electroacupuncture — The primary acupoints selected were the affected side's Sibai (ST2), Xiaguan (ST7), and Dicang (ST4). Based on the affected nerve branch, additional acupoints were chosen: for the ophthalmic branch, Tongziliao (GB1); for the maxillary branch, Quanliao (SI18); and for the mandibular branch, Jiache (ST6). Distal acupoints included bilateral Hegu (LI4) and Waiguan (SJ5). Electroacupuncture was applied based on the affected nerve branch. For the ophthalmic branch, the local acupoints selected were Xiaguan + Tongziliao; for the maxillary branch, Xiaguan + Quanliao; and for the mandibular branch, Xiaguan + Jiache. The distal acupoints selected were Hegu + Waiguan. A sparse-dense wave, 2/100Hz, was used, with a treatment duration of 60 minutes. The intensity of the electrical current was adjusted according to the patient's tolerance. Acupuncture treatment is administered in 5 consecutive days as one course, with a 2-day break between courses. A total of 2 courses are conducted.
  Arms: EA+placebo group

SUMMARY:
Trigeminal neuralgia (TN), characterized by its refractory nature and recurrence, frequently leads to anxiety, depression, and insomnia, thereby significantly diminishing patients' quality of life and potentially inducing self-harm. Carbamazepine (CBZ) is the first-line medication for TN, yet it presents adverse effects such as addiction and the absence of analgesic effects upon cessation. Acupuncture, particularly electroacupuncture（EA）, has demonstrated efficacy in TN treatment, although its therapeutic outcomes are influenced by various factors. Consequently, this study aims to evaluate the clinical efficacy of EA for TN and its potential as an alternative to CBZ treatment.

DETAILED DESCRIPTION:
This study will enroll a total of 126 patients with TN who meet the inclusion criteria. Participants will be randomized in a 1:1 ratio to either the EA plus placebo group or the sham EA plus CBZ group. This study aims to investigate the clinical efficacy of EA for TN and to determine if EA offers a viable therapeutic alternative for TN management.

ELIGIBILITY:
Diagnostic Criteria

Diagnosis was based on the criteria for trigeminal neuralgia (TN) as defined in the third edition of the International Classification of Headache Disorders (ICHD-3) published by the International Headache Society (IHS) in 2018. The diagnostic criteria included:

1. recurrent unilateral facial pain occurring in the distribution of one or more divisions of the trigeminal nerve, without radiation outside the trigeminal territory, and meeting criteria (2) and (3);
2. pain presenting with all of the following characteristics:

   ① paroxysmal attacks lasting from a few seconds to 2 minutes;

   ② severe intensity;
   * electric shock-like, stabbing, or sharp quality;
3. pain triggered by innocuous stimuli within the affected trigeminal distribution;
4. exclusion of other facial pain disorders classified in ICHD-3.

   Inclusion Criteria

   All of the following criteria had to be met for study enrollment:
   * fulfillment of the TN diagnostic criteria as stated above;

     * age between 18 and 80 years, inclusive, irrespective of sex;

       * receiving a stable daily dose of carbamazepine (200-400 mg); ④ consciousness clear, with intact pain perception and discrimination, and able to communicate effectively; ⑤ voluntary participation with written informed consent provided by the patient or their legal guardian/authorized representative.

   Exclusion Criteria

   Participants were excluded if they met any of the following:
   * comorbid epilepsy, head injury, or other relevant neurological disorders;

     * significant impairment of cardiac, hepatic, or renal function;

       * cognitive dysfunction, aphasia, psychiatric conditions, or inability to cooperate with treatment;

         * poorly controlled hypertension or hyperglycemia;

           ⑤ recent diagnosis of severe anxiety or depression;

           ⑥ pregnancy or lactation;

           ⑦ presence of a cardiac pacemaker or other contraindications to electroacupuncture therapy;

           ⑧ current participation in another clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
VAS Response Rate | Baseline, the end of the 2-week treatment.
  The proportion of patients with a reduction in VAS score of ≥50% from baseline at the end of the 2-week treatment.

SECONDARY OUTCOMES:
Changes in Visual Analog Scale (VAS) scores | At baseline, and at the end of weeks 2, 4, and 8.
  Changes in VAS scores from baseline at weeks 2, 4, and 8.
Pain Diary Card | Daily from baseline through the end of week 8.
  Patients were required to complete a 24-hour pain diary card daily. The diary included the following items: (a) the daily frequency of pain episodes (including both spontaneous and triggered episodes); (b) triggering factors; (c) the average pain intensity over the past 24 hours (assessed using a visual analog scale [VAS]); (d) the highest pain intensity over the past 24 hours (VAS); (e) adverse events within the past 24 hours (including those related to medication or acupuncture); and (f) whether any pain relief methods outside the study protocol were used, and if so, specify the method.
Changes in the Patient global impression of change （PGIC） | At baseline, and at the end of weeks 2, 4, and 8.
  The Patient Global Impression of Change (PGIC) scale is a patient-reported outcome measure used to dynamically monitor the trajectory of health status. This scale employs a seven-point Likert scale (1=very much worse to 7=very much better) to assess the impact of therapeutic interventions on an individual's functional status. Treatment efficacy is categorized into three levels: ① disease progression (scores 0-3) indicates a worsening of symptoms; ② functional stability (score 4) suggests no significant change in symptoms; and ③ clinical improvement (scores 5-7) represents a marked reduction in symptoms. This subjective assessment tool, through longitudinal comparison with baseline data, provides a direct reflection of the patient's perceived treatment benefit.
Changes in the Brief pain inventory-facial scale （BPI-Facial） | At baseline, and at the end of weeks 2, 4, and 8.
  The Brief Pain Inventory-Facial Scale (BPI-Facial) is designed to establish a three-dimensional assessment system: ① Pain intensity dimension (4 items) quantifies the frequency and severity of pain; ② Daily function dimension (7 items) assesses the impact of pain on basic life activities (including specific emotional states); ③ Facial function dimension (7 items) detects the degree of limitation in specific facial activities. Eighteen standardized items, measured from multiple perspectives, can systematically evaluate pain-related physiological, psychological, and social functional changes, providing multidimensional data support for efficacy determination.
Changes in the Short-Form McGill Pain Questionnaire （SF-MPQ） | At baseline, and at the end of weeks 2, 4, and 8.
  The Short-Form McGill Pain Questionnaire (SF-MPQ) innovatively integrates qualitative and quantitative analyses of neuropathic pain. This involves: (1) Pain quality assessment: Utilizing 11 sensory descriptors (e.g., pricking, burning) and 4 affective descriptors (e.g., annoying, fearful), a 0-3 intensity rating system is established, synthesizing a Pain Rating Index (PRI = sensory score + affective score); (2) Pain intensity assessment: Employing a Visual Analog Scale (VAS) and the Present Pain Intensity index (PPI) for supplementary quantification. This scale significantly enhances clinical applicability while maintaining assessment validity, and has become a gold standard for neuropathic pain assessment.
Changes in the The Self-Rating Anxiety Scale (SAS) | At baseline, and at the end of weeks 2, 4, and 8.
  In assessing anxiety via the Self-Rating Anxiety Scale (SAS), scoring yields two key metrics: the raw sum score (X) and the derived standard score (Y). The latter is calculated as the integer portion of 1.25X, with truncation applied. Per Chinese norms, a standard score (Y) of 50 serves as the threshold for clinical anxiety, with severity stratified as mild (50-59), moderate (60-69), or severe (≥70).
Changes in the Self-Rating Depression Scale (SDS) | At baseline, and at the end of weeks 2, 4, and 8.
  The Self-Rating Depression Scale (SDS) is a brief, self-rated instrument for assessing depressive symptomatology. The total raw score (X) is derived by summing all item responses, which is then converted to a standard score (Y) by multiplying by 1.25 and truncating to an integer. Based on Chinese normative data, a standard score cutoff of 53 is adopted, with scores of 53-62, 63-72, and ≥73 indicating mild, moderate, and severe depression, respectively.